CLINICAL TRIAL: NCT01925690
Title: Development of a Motivational Intervention to Improve Treatment Adherence in MS
Acronym: MIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Jared Bruce, Associate Professor of Psychology, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0033769; National MS Society (Other Grant/Funding Number: National MS Society)
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Disease modifying medication; Relapsing-Remitting MS; Motivational Interviewing; Telephone Counseling
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Education (Active Comparator): Patients receive a brief educational packet along with treatment as usual
  Interventions: Behavioral: Brief Education
- MI-CBT Treatment (Experimental): Patients receive five 20 minute phone sessions of motivational interviewing/cognitive behavioral therapy weekly along with a brief educational packet.
  Interventions: Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy; Behavioral: Brief Education

INTERVENTIONS:
Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy — A telephone based talk therapy discussing pros and cons of medication use in MS.
  Arms: MI-CBT Treatment
Behavioral: Brief Education — Give patients a pamphlet discussing pros and cons of disease modifying therapies

SUMMARY:
As many as 50% of MS patients prematurely discontinue their disease modifying medications. For this study, we will develop a telephone-based talk therapy intervention and then conduct a randomized controlled trial. Patients will be assigned to either 5 weekly 20 minute telephone sessions of psychotherapy or a brief education control condition. We hypothesize that patients undergoing phone therapy will be more likely to indicate they are interested in resuming taking disease modifying medications than patients given brief education and treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remitting MS based on established guidelines
* Previously discontinued recommended therapy
* Provider recommendation for DMT re-initiation
* At least 18 years of age
* Access to a telephone
* English speaking

Exclusion Criteria:

* Diagnosis other than relapsing remitting MS
* Provider does not recommend DMT re-initiation
* Pregnant or breastfeeding (females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adherence Treatment Survey | 10 weeks after enrollment
  Whether the patient indicates if he/she decided to re-initiate disease modifying therapies on a "yes"/"no" question.

SECONDARY OUTCOMES:
Adherence Treatment Survey | 10 weeks after enrollment
  Whether the patient reports that he/she plans to discuss disease modifying therapies with a care provider on a "yes"/"no" question.
Adherence Treatment Survey | 5 weeks after enrollment
  Whether the patient reports that he/she plans to discuss disease modifying therapies with a care provider on a "yes"/"no" question.
Adherence Treatment Survey | 5 weeks after enrollment
  Whether the patient indicates if he/she decided to re-initiate disease modifying therapies on a "yes"/"no" question.

OTHER OUTCOMES:
Motivation/Readiness Questionnaire | 10 weeks post-enrollment
  Whether there is increased self-reported motivation to take disease modifying therapies on a 1-10 likert-type scale.
Motivation/Readiness Questionnaire | 5 weeks post-enrollment
  Whether there is an increase in self-reported motivation to take disease modifying therapies on a 1-10 likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jared M Bruce, Ph.D., Principal Investigator — University of Missouri, Kansas City
Locations (2):
- United States (2):
  - University of Missouri-Kansas City, Kansas City, Missouri
  - Kessler Rehabillitation Institute, West Orange, New Jersey

REFERENCES:
- [Derived] Bruce J, Bruce A, Lynch S, Strober L, O'Bryan S, Sobotka D, Thelen J, Ness A, Glusman M, Goggin K, Bradley-Ewing A, Catley D. A pilot study to improve adherence among MS patients who discontinue treatment against medical advice. J Behav Med. 2016 Apr;39(2):276-87. doi: 10.1007/s10865-015-9694-6. Epub 2015 Nov 12. PMID 26563147
- See also: Clinical Neuropsychology Lab Research — https://sites.google.com/site/clinicalneuropsychologylab/contact-us